CLINICAL TRIAL: NCT02417597
Title: Safety and Immunogenicity Study of the Recombinant Hepatitis E Vaccine(Escherichia Coli) in Healthy Volunteers Aged Over 65 Years
Brief Title: A Phase Ⅳ Clinical Trial of the Recombinant Hepatitis E Vaccine (Escherichia Coli)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xiamen Innovax Biotech Co., Ltd (Industry)
Collaborators: Xiamen University (Other); Beijing Wantai Biological Pharmacy Enterprise Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-HE-006
Record Dates: First submitted 2015-04-11; First posted 2015-04-15 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2015-10

CONDITIONS: Hepatitis E
Keywords: hepatitis E
MeSH Terms: conditions — Hepatitis E | interventions — hecolin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Experimental Group (Experimental): Participants in this arm are aged over 65 years and would receive three doses of Recombinant Hepatitis E Vaccine (Escherichia Coli)(Hecolin®) at o,1,6 month.
  Interventions: Biological: Recombinant Hepatitis E Vaccine (Escherichia Coli)
- Immunogenicity Control Group (Active Comparator): Participants in this arm are aged beteen 18-65 years and would receive three doses of Recombinant Hepatitis E Vaccine (Escherichia Coli)(Hecolin®) at o,1,6 month.
  Interventions: Biological: Recombinant Hepatitis E Vaccine (Escherichia Coli)
- Safety Control Group (No Intervention): Participants in this arm are aged over 65 years.

INTERVENTIONS:
Biological: Recombinant Hepatitis E Vaccine (Escherichia Coli) — Participants would intramuscularly receive 3 doses of Recombinant Hepatitis E Vaccine (Escherichia Coli) at 0, 1, 6 month.
  Other Names: Hecolin®
  Arms: Experimental Group; Immunogenicity Control Group

SUMMARY:
This phase IV clinical study was designed to evaluate the safety and immunogenicity of the recombinant Hepatitis E vaccine(Hecolin®), manufactured by Xiamen Innovax Biotech CO., LTD., in healthy volunteers aged over 65 years of age at enrollment. The study volunteers will receive the 3 doses of Hecolin® administered intramuscularly according to a 0-1-6 month schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy people aged over 18 years old on the day of enrollment
2. Axillary temperature is below than 37.0 ℃
3. Blood pressure is not higher than 160/100 mmHg (with or without any medicine)
4. Judged as healthy and eligible for vaccination by the investigators through a self-reported medical history and some physical examinations.
5. Able to understand this study information and willing to comply with all study requirements.
6. Willing to participate in this study and sign informed consent form.

Exclusion Criteria:

1. Participated in any other clinical trial during the study period.
2. Use of any investigational product or non-registered product (drug or vaccine) within 30 days preceding the first dose of the study vaccine or plan to use during the study period.
3. Received immunosuppressed, immunoregulation therapy or corticosteroid systemic therapy for more than 14 days in the 6 months before entry, except local treatment.
4. Administration of any immunoglobulin or blood products within 3 months preceding the first dose of the study vaccine,or plan to use during the study period.
5. Administration of any inactivated vaccines within 14 days preceding the first dose of the study or attenuated live vaccines within 21 days preceding the first dose of the study.
6. Had a fever (axillary temperature over 38°C) within 3 days or acute illness requiring systemic antibiotics or antiviral treatment within 5 days before vaccination.
7. Immunodeficiency (such as HIV carriers), primary disease of important organs, malignant tumor, .or any immune disease (such as systemic lupus erythematosus, arthritis pauperum, splenectomy or functional asplenia or other disease which might affect immune response).
8. History of allergic disease or history of serious adverse events occurring after vaccination, i.e., allergy,urticaria, dyspnea, angioneurotic edema or abdominal pain.
9. Pregnant or breastfeeding
10. Allergic history to any component of this vaccine.
11. Other medical, psychological, social or occupational factors that, according to the investigators' judgment,might affect the individual's ability to obey the protocol or sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2015-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Adverse reactions/events | up to 10 months
  Measure solicited local adverse reactions within 7 days after each vaccination; Measure solicited systematic adverse reactions within 7 days after each vaccination; Measure unsolicited adverse reactions within 30 days after vaccination; Measure serious adverse events occurred throughout the study

SECONDARY OUTCOMES:
Anti-HEV antibody | 7 months
  Measure anti-HEV antibody in serum samples at 7 month to evaluate the immunogenicity of the Hepatitis E vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiping Chen, Principal Investigator — Zhejiang Provincial Center for Disease Control and Prevention
Locations (1):
- Kaihua Center for Disease Control and Prevention, Quzhou, Zhejiang, China

REFERENCES:
- [Derived] Yu XY, Chen ZP, Wang SY, Pan HR, Wang ZF, Zhang QF, Shen LZ, Zheng XP, Yan CF, Lu M, Chen B, Zheng Y, Zhang J, Lv HK, Huang SJ. Safety and immunogenicity of hepatitis E vaccine in elderly people older than 65 years. Vaccine. 2019 Jul 26;37(32):4581-4586. doi: 10.1016/j.vaccine.2019.04.006. Epub 2019 Jun 28. PMID 31262585